CLINICAL TRIAL: NCT00527761
Title: Phase I Study of TTC (Taxotere/Temodar/Cisplatin) in Metastatic Melanoma Patients
Brief Title: Taxotere/Temodar/Cisplatin Study in Melanoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-1037
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Metastatic Melanoma
Keywords: Metastatic Melanoma; Temozolomide; Temodar; Taxotere; Cisplatin; TTC
MeSH Terms: conditions — Melanoma | interventions — Cisplatin; Docetaxel; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temozolomide, Docetaxel + Cisplatin (Experimental)
  Interventions: Drug: Cisplatin; Drug: Docetaxel; Drug: Temodar

INTERVENTIONS:
Drug: Cisplatin — 20 mg in 500 ml of normal saline by vein over 60 minutes daily for 4 days starting on day 1 of chemotherapy.
  Other Names: Platinol-AQ; Platinol; CDDP
Drug: Docetaxel — Starting dose 20 mg by vein over 1 hour, once a week, for three weeks (on Days 1, 8, and 15).
  Other Names: Taxotere
Drug: Temodar — 150 mg by mouth (PO) on Days 1 - 5.
  Other Names: Temozolomide

SUMMARY:
Primary Objective:

1. To determine the maximum tolerated dose of chemotherapy using Taxotere, Temodar, Cisplatin (TTC) in patients with metastatic melanoma.

Secondary Objectives:

1. To determine the toxicity of chemotherapy using Taxotere, Temodar, Cisplatin (TTC) in patients with metastatic melanoma
2. To determine the response rate of induction chemotherapy using Taxotere, Temodar, Cisplatin (TTC) in patients with metastatic melanoma.

DETAILED DESCRIPTION:
Temozolomide, docetaxel, and cisplatin are "chemotherapy" drugs, known to kill tumor cells by interfering with the important structures in these cells to grow and divide. Each of these drugs has been used separately for melanoma treatment. These 3 drugs have not been used in combination.

Before you can start treatment on the study, you will have what are called "screening tests". These tests will help the doctor decide if you are eligible to take part in the study. You will have a complete medical history and physical exam, including routine blood tests (less than 3 tablespoons). You will have an electrocardiogram (EKG - test to measure the electrical activity of the heart), a chest x-ray, and CT scans of the chest and abdomen. You will have a MRI or CT scan of brain will as well. Depending on the location of melanoma, CT scans of the head and neck or pelvis and/or a bone scan may be taken. Photographs of the tumor may be taken if the tumors are located on the surface of the skin. Women who are able to have children must have a negative blood pregnancy test.

If you are found to be eligible, you will receive temozolomide, cisplatin, and docetaxel. The doses of temozolomide and cisplatin will be fixed for all groups. The dose of docetaxel will be changed between patient groups until the highest safe dose is found Between 3 and 6 patients will be enrolled in each group. Docetaxel will be given by vein over 1 hour, once a week, for three weeks (on Days 1, 8, and 15). This will be followed by one week of rest. These 3 weeks of treatment and 1 week or rest make up 1 cycle. Cisplatin will be given by vein once a day for four days in a row (Days 1, 2, 3 and 4) over 2 hours each cycle. Temozolomide will be taken by mouth for five days in a row (Days 1, 2, 3, 4 and 5) of each cycle. The number of temozolomide pills that you take will be based on your height and weight. Temozolomide must be taken on an empty stomach (at least 2 hours before or after meals).

For your comfort in receiving cisplatin and docetaxel by vein, your doctor may recommend a catheter. A catheter is a plastic tube that is inserted into a vein in one of your arms or into the vein that runs underneath the collar bone, and then threaded into the central vein in the upper part of the chest.

The first dose of docetaxel and all of the cisplatin doses must be given at M.D. Anderson on an outpatient basis. All of the temozolomide doses can be taken at home and the Day 8 and Day 15 doses of docetaxel can be taken at a local clinic.

You may receive granulocyte colony-stimulating factor (G-CSF) to help the body produce new blood cells. G-CSF would be given as an injection under the skin on Days 9-13 of each cycle (except the first cycle).

During the study, you will have a complete physical exam every 4 weeks. Blood samples (1 tablespoon or less) will be taken weekly to monitor the blood counts and liver functions. A chest x-ray and CT scans of the chest and abdomen with or without head and neck and pelvis will be done every 2 cycles (8 weeks). A MRI or CT scan of the brain as well as photographs may also be taken every 2 cycles during the study. For patients who have significant tumor shrinkage with the treatment, these imaging studies may be repeated in 4 weeks.

All participants can receive at least 6 cycles of treatment. If your tumor continues to shrink after the end of 6 cycles, you may be eligible to receive further treatment at the discretion of the study chair. You may be taken off study early, if your disease gets worse or intolerable side effects occur.

You will have one last "follow-up" visit once you are taken off study. At this visit you will have a complete physical exam and blood samples (1 tablespoon) for routine tests will be taken. You will have a chest x-ray and CT scans of the chest and abdomen, with or without head and neck and pelvis, and with or without a MRI of brain at this visit as well.

This is an investigational study. The FDA has approved all of the drugs in this study, and they are commercially available. However, their use together in this study is experimental. Up to 30 patients will take part in this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 or older with histologically documented diagnosis of advanced/inoperable melanoma are eligible.
2. Patients must have measurable metastatic melanoma lesion(s), and at least 1 lesion must be greater then or equal 10 mm in a greatest diameter by spiral CT scan (or greater then or equal to 20 mm by a conventional non-spiral CT scan) to assess response. Cutaneous lesions may be 10 mm or larger in a greatest diameter.
3. Patients with less than or equal to grade 1 peripheral neuropathy at the time of enrollment.
4. Patients with controlled, asymptomatic brain metastases will be eligible. There should not be any evidence of progression in the brain metastases for at least 3 months after the complete surgical resection/stereotactic radiosurgery and/or a whole brain radiation therapy. Patients who are taking steroidal or anticonvulsant drug(s) for brain metastasis at the time of registration will not be eligible.
5. Zubrod performance status of 0-2.
6. ANC greater than or equal to 1,500/mm3 and a platelet count greater than or equal to 100,000/mm3.
7. Serum creatinine less than or equal to 1.5 mg/dl
8. Serum bilirubin level of less than or equal to 1.0 mg/dl (or up to institutional upper limit of normal (ULN))
9. Serum transaminase (ALT and AST) less than or equal to 125 IU/l (or up to 2.5 x institutional ULN) if alkaline phosphatase is less than or equal to 130 IU/l (or institutional ULN), or alkaline phosphatase less than or equal to 500 IU/l (or up to 4 x ULN) if transaminases are less than or equal to 50 IU/l (or institutional ULN).
10. No evidence of significant cardiac or pulmonary dysfunction.
11. Patient must have a hemoglobin greater than or equal to 9 gm/dl (this may be achieved by transfusion if needed) obtained within 14 days prior to registration. If a patient receives PRBC transfusion to achieve a hemoglobin level of greater than or equal to 9 gm/dl, the hemoglobin level needs to be stable (no drop by more than 1 gm/dl from the post-transfusion hemoglobin level) for at least 1 week.
12. Women of childbearing potential must have a negative pregnancy test and may not be breastfeeding.
13. Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
14. All patients must be informed of the investigational nature of this study and must sign and give written informed consent for treatment and in accordance with institutional and federal guidelines.

Exclusion Criteria:

1. A prior exposure to all 3 drugs: taxanes, Temodar and platinum.
2. A history of severe hypersensitivity reaction to drugs formulated with polysorbate 80.
3. Any anti-cancer therapy within 28 days prior to enrollment.
4. If a target lesion has been previously embolized, perfused or irradiated, there must be objective evidence of progression before start of therapy to be considered for response assessment.
5. Uncontrolled brain metastases. Patient who is symptomatic from brain metastases or who takes steroidal or anticonvulsant drug for the management of brain metastases will be ineligible. Central nervous system involvement by melanoma either as spinal cord compression or leptomeningeal disease will also be excluded.
6. Patients with significant cardiac illness such as symptomatic coronary artery disease or previous history of myocardial infarction, impaired left ventricle function (EF less than 55%) on account of any organic disease such as hypertension or valvular heart disease or serious uncontrolled cardiac arrhythmias despite therapy.
7. Patients with significant impairment of pulmonary function on account of chronic bronchitis or chronic obstructive pulmonary disease (COPD) which has resulted in impairment of vital capacity or FEV1 to less than 75% of predicted normal values.
8. Symptomatic effusions on account of pleural, pericardial or peritoneal metastasis of melanoma.
9. No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, surgically treated Stage I or II cancer from which the patient is currently in complete remission (at least for 5 years), or any other cancer from which the patient has been disease-free for 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 4 week cycles

CONTACTS AND LOCATIONS:
Overall Officials: Kevin B. Kim, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org